CLINICAL TRIAL: NCT07368270
Title: A Prospective, Open-label and Single-arm Study of Anti-PD1 Armored CD19 CAR-T Cells in Adult Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Safety and Efficacy Study of Anti-PD1 Armored CD19 CAR-T Cells in Adult Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-RD09-02
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD1 armored CD19 CAR-T cells treatment arm (Experimental): Subjects will be administrated with Anti-PD1 armored CD19 CAR-T cells after lymphocyte depletion by fludarabine and cyclophosphamide.
  Interventions: Biological: Anti-PD1 armored CD19 CAR-T cells

INTERVENTIONS:
Biological: Anti-PD1 armored CD19 CAR-T cells — Anti-PD1 armored CD19 CAR-T cells, single intravenous infusion

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of anti-PD1 armored CD19 CAR-T Cells in adult subjects with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm clinical study to evaluate the safety, tolerability of anti-PD1 armored CD19 CAR-T Cells in adult subjects with relapsed or refractory diffuse large B-cell lymphoma (r/r DLBCL).The study plans to explore across three dose levels (1.00 × 10^6, 3.00 × 10^6, 9.00 × 10^6 CAR+ T cells/kg), and 6.00×10^8 CAR+T cells as maximum dose, aiming to evaluate the safety, tolerability of anti-PD1 armored CD19 CAR-T Cells in r/r DLBCL, explore Maximum Tolerated Dose (MTD) and determine the recommended dose for Phase II. Besides, efficacy, pharmacokinetics and persistence profile of CAR-T cells are also study objectives.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily participate in clinical research and sign informed consent.
* 2. Adult subjects (age ≥18 ) with relapsed or refractory diffuse large B-cell lymphoma: a) failure to achieve CR after 6 cycles, or PR after 3 cycles, of first-line therapy, or achieve CR after first-line therapy but relapse within 12 months; b) achieve CR after systemic treatment, but are refractory or relapsed, and no plan to transplant, or prepare for transplantation but cannot meet transplantation criteria after second-line therapy; c) not achieve CR after at least two courses of second-line treatment (including autologous stem cell transplantation).
* 3. Expected survival ≥ 3 months.
* 4. At least one measurable lesion as per revised IWG response criteria for malignant lymphom (2014 Lugano criteria).
* 5. CD19 positive expression are detected on tumor cells of subjects by flow cytometry or immunohistochemistry.
* 6. ECOG score ≤ 2.
* 7. Subjects with adequate organ functions prior to enrollment, meet the following laboratory values:
* Renal function: serum creatinine ≤ 1.5 × ULN or estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m².
* Hepatic function: Serum alanine aminotransferase (ALT) ≤ 5 × age-specific ULN and total bilirubin ≤ 2.0 mg/dL, except in subjects with Gilbert-Meulengracht syndrome. If total bilirubin ≤ 3.0 × ULN and direct bilirubin ≤ 1.5 × ULN, subjects with Gilbert-Meulengracht syndrome are included.
* Pulmonary reserve: ≤ Grade 1 dyspnea and oxygen saturation >95% on room air.
* 8. Stable hemodynamics and left ventricular ejection fraction (LVEF) ≥ 45 % assessed by echocardiography or multi-gated radionuclide angiography (MUGA).
* 9. Adequate bone-marrow reserve without blood transfusion as defined by:
* Absolute neutrophil count (ANC) ≥ 1 x 10^9/L.
* Absolute lymphocyte count (ALC) ≥ 0.1 x 10^9/L.
* Platelets ≥ 50 x 10^9/L.
* Hemoglobin >80g/L.
* 10. In the investigator's judgment, subjects' general condition and all biochemical values are either normal or sufficiently compensated to receive lymphodepletion and CAR-T cell therapy.

Exclusion Criteria:

* 1. Women who are pregnant or breastfeeding, or planned pregnancy within 6 months.
* 2. Infectious disease(HIV, Active Tuberculosis ect.).
* 3. Active infection: hepatitis B, hepatitis C.
* 4. Abnormal vital signs or refuse to receive examination.
* 5. Subjects with psychiatric or psychological disorders are unable to complete treatment or efficacy assessment.
* 6.History of severe hypersensitivity or known hypersensitivity to IL-2.
* 7. Systemic or local severe infection requiring antimicrobial therapy.
* 8. Significant dysfunction of vital organs (heart, lung, brain, kidney, etc.), or in the investigator's judgment, subjects are unable to be enrolled with any other condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 1 month after injection
  Dose-limiting toxicity for each subject
AE/SAE | 1 month, 3 months, 6 months, 12 months after injection
  Incidence and severity of adverse events (AE), and serious adverse event (SAE)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 month, 3 months, 6 months, 9 months, 12 months after injection
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients
Overall survival (OS) | 1 month, 3 months, 6 months, 9 months, 12 months after injection
  Defined as the time from the date of first infusion to death due to any cause
Duration of response (DOR) | 1 month, 3 months, 6 months, 9 months, 12 months after injection
  The time from the date of first response (PR or better) to the date of disease progression after infusion
Progression-free survival (PFS) | 1 month, 3 months, 6 months, 9 months, 12 months after injection
  The time from first infusion to the date of progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hongci Hematology Hospital, Suzhou, China

IPD SHARING:
Plan to Share IPD: No